CLINICAL TRIAL: NCT02452567
Title: Effect of Moderate Weight Loss in Metabolically Abnormal Lean Subjects
Acronym: MAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting participants that met the inclusion criteria
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201501010
Record Dates: First submitted 2015-04-15; First posted 2015-05-22 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metabolically abnormal lean (Experimental): Moderate (8-10%) diet-induced weight loss.
  Interventions: Other: Moderate (8-10%) diet-induced weight loss

INTERVENTIONS:
Other: Moderate (8-10%) diet-induced weight loss — MAL participants will meet with the study dietitian to lose ~8-10% of their body weight through diet-intervention.

SUMMARY:
Obesity is associated with a constellation of cardiometabolic abnormalities (including insulin resistance, elevated blood pressure and dyslipidemia) that are risk factors for diabetes and cardiovascular disease. Weight loss can improve all of the cardiometabolic abnormalities associated with obesity. Up to ~25% of lean people (Body Mass Index [BMI] 18.5-24.9 kg/m²) have many of the cardiometabolic abnormalities associated with obesity and are referred to as metabolically abnormal lean (MAL) people. However, the MAL phenotype is not well characterized, and it is unclear whether weight loss has beneficial metabolic effects in already lean people. Accordingly, the goal of this study is to: 1) carefully phenotype MAL people and 2) evaluate the effect of moderate (8-10%) diet-induced weight loss in MAL people. This will be investigated in 15 MAL (defined as having 2 or more of the following: intrahepatic triglyceride (IHTG) content ≥5.6%, glycated hemoglobin ≥5.7%, fasting plasma glucose concentration ≥100 mg/dl, 2-hr oral glucose tolerance test (OGTT) plasma glucose concentration ≥140 mg/dl, homeostatic model assessment of insulin resistance (HOMA-IR) ≥ 2.5) men and women. Only lean people who have a BMI ≥21.0 but <25.0 kg/m² will be asked to lose weight to avoid the risk that participants become underweight (BMI <18.5 kg/m²) during weight loss therapy.

ELIGIBILITY:
Inclusion Criteria:

* BMI 21.0-24.9 kg/m²
* Weight stable (+/- 2% for at least 3 months before enrollment)
* Two or more of the following: IHTG content ≥5.6%, HOMA- IR index ≥ 2.5, HbA1C ≥ 5.7%, 2-hr OGTT plasma glucose concentration ≥ 140 mg/dl, fasting plasma glucose concentration ≥ 100 mg/dl.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Evidence of significant organ system dysfunction or disease (e.g., diabetes, chronic kidney disease, advanced heart disease, etc.)
* Men who consume >21 units (e.g., glass of wine or bottle of beer) of alcohol per week and women who consume >14 units of alcohol per week
* Use of dietary supplements or medications known to affect metabolism
* Eating disorder (assessed by using the Eating Disorder Examination Questionnaire [EDE-Q])
* Participation in structured endurance or resistance exercise program >150 min/week
* Use of tobacco products
* Unable or unwilling to follow the study protocol or the research team believes that for any reason the volunteer is not an appropriate candidate for this study, including non-compliance with screening appointments or previous appointments/contact arrangements
* Individuals that take Coumadin or similar anticoagulants
* Use of antibiotics in last 60 days
* Previous bariatric surgery
* Cancer or cancer that has been in remission for <5 years
* Major psychiatric illness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity as assessed by the hyperinsulinemic-euglycemic clamp technique | An average of 6-8 months from baseline testing to 8-10% weight loss
  Evaluate insulin sensitivity through the hyperinsulinemic-euglycemic clamp procedure.

SECONDARY OUTCOMES:
Change in Beta-Cell function | An average of 6-8 months from baseline testing to 8-10% weight loss
  Administer 3 hour oral glucose tolerance test before and after weight loss to determine the effects of weight loss on beta cell function
Change in fat mass and fat free mass as assessed by dual-energy x-ray absorptiometry (DXA) | An average of 6-8 months from baseline testing to 8-10% weight loss
Change in intra-abdominal adipose tissue volume as assessed by magnetic resonance imagining. | An average of 6-8 months from baseline testing to 8-10% weight loss
  Inta-abdominal adipose tissue volume will be assessed before and after weight loss to determine the effects of weight loss
Change in plasma lipid profile as assessed by the complete metabolic panel and lipid panel. | An average of 6-8 months from baseline testing to 8-10% weight loss
  Blood will be drawn for the complete metabolic panel and lipid panel before and after weight loss
Change in markers of inflammation in plasma and adipose tissue as assessed from samples obtained during the hyperinsulinemic-euglycemic clamp procedure with adipose tissue biopsies | An average of 6-8 months from baseline testing to 8-10% weight loss
  Plasma samples and adipose tissue biopsies will be obtained during the hyperinsulinemic-euglycemic clamp procedure before and after weight loss
Change in cellular factors involved in mediating insulin action in muscle and adipose tissue as assessed by muscle and adipose tissue biopsies obtained during the hyperinsulinemic-euglycemic clamp procedure | An average of 6-8 months from baseline testing to 8-10% weight loss
  Muscle and adipose tissue biopsy samples will be obtained during the hyperinsulinemic-euglycemic clamp procedure before and after weight loss
Modification of gut microbiota | An average of 6-8 months from baseline testing to 8-10% weight loss
  Monthly stool collection will be used to assess the composition of the gut microbiota, meta-transcriptome (bacterial RNA sequencing to determine what proteins can be made by the microbiota), and the meta-metabolome (metabolites made by the microbiota).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States